CLINICAL TRIAL: NCT01315860
Title: Association of Biomechanical Changes and Weight Gain Throughout Pregnancy
Status: Completed | Type: Observational
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Natalie Wessel, OMS III, Nova Southeastern University
Other Study IDs: 01111110Exp.
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Low Back Pain; Pregnancy
Keywords: Low Back Pain; Pregnancy; Biomechanics
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnant Females: Pregnant females in their second or third trimester that meet the inclusion and exclusion criteria.
  Interventions: Other: Postural Analysis

INTERVENTIONS:
Other: Postural Analysis — Measure the subject's weight, sway rate and shift of center of gravity on a postural scale for 15 seconds. Measure lumbosacral angle with an inclinometer.

SUMMARY:
Low back and posterior pelvic pain are common in pregnant females. Previous studies have demonstrated disability and it is estimated that all women experience some degree of musculoskeletal discomfort during pregnancy. Borg-Stein et. al. found 25% of pregnant females have temporarily disabling symptoms.

There is demonstrated controversy over the mechanism of low back pain in pregnancy. The biomechanical theory implies that the enlarging uterus causes the maternal center of gravity to move anteriorly causing stress on the low back. Jensen et. al. demonstrated that weight gain correlated with biomechanical changes. The changes were measured by weight gain in segmental regions of the body and in principal moments of inertia from the sit to stand movement. Literature does not demonstrate a specific correlation between weight gain and the biomechanical changes of sway rate, lumbosacral angle and center of gravity. These three measurements may have a correlating effect on the underlying cause of low back pain in pregnant women.

This study aims to determine the correlation between weight gain of pregnant females and the biomechanical changes of sway rate, lumbosacral angle and center of gravity. The change in weight over the last two trimesters will be correlated with the sway rate, lumbosacral angle and center of gravity. The degree of symptomatic low back pain as measured by the Oswestry Low Back Pain Scale will also be correlated with the sway rate, lumbosacral angle and center of gravity.

DETAILED DESCRIPTION:
The principal investigator will recruit subjects at the yoga studio and one of the investigators and the research assistant will recruit subjects at the NSU clinic. Potential subjects will go through a short verbal pre-screening to ensure they fit the inclusion and exclusion criteria. Subjects that fit this criteria will read and sign the consent form. The PI and research assistant will answer any questions about the study prior to the subject giving consent.

Then the subject's initial weight will be measured on the postural scale and documented. Change in weight is the dependent variable in this study. The following independent variables will be measured: lumbosacral angle, sway rate and shift of weight posteriorly. The lumbosacral angle will be measured by a digital inclinometer. The lumbosacral angle is measured between the plane of the superior surface of S1 to the horizontal plane. Saur et. al., demonstrated that the inclinometer technique for lumbosacral angle has established validity and reliability in comparison to radiographic x-rays. Comparison of radiographic and inclinometer technique is clinically suitable for measuring lumbar position. Keeley et. al. reported high correlation coefficients for interrater reliability with the inclinometer technique on patients with chronic low back pain.

The additional measurements of sway rate and center of gravity will be measured by the postural analyzer. The quadruple scale that will be used in this study is based on four digital force plates with computer communication operated by software enabling test analysis. The quadruple scale will provide numeric and graphic data on total weight, weight distribution (kg. or lb.), percentage weight difference, sway rate and an estimate of the location and deviation of the subject's center of mass. All data will be recorded and saved.

Following those measurements, the subject will be asked to complete the Oswestry Low Back Pain Scale. The Oswestry Low Back Pain Scale is a suitable questionnaire for an English-speaking population and to enquire about areas of functioning specifically relevant to low back pain sufferers, such as lifting, walking, sitting, standing, sleeping and socializing. Fisher et. al. demonstrated that the Oswestry Low Back Pain Scale is an acceptable instrument for back pain patients with evidence of criterion-related validity, factorial validity and moderately high internal consistency. It has good face validity for the patients. According to Fisher et. al., the Oswestry Scale can be recommended as a relevant measure of disability with evidence of validity, reliability and sensitivity to change for both clinical and research purposes.

The total amount of time needed to complete the measurements and the Oswestry Low Back Pain Scale should take 15 minutes. Biweekly, willing participants will be recruited and previous participants will be continually measured for weight, lumbosacral angle, sway rate and deviation of the subject's center of mass.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients in their second or third trimester who are patients at NSU Ob/Gyn clinic or prenatal yoga students at Red Pearl Yoga Studio who are willing to participate in the study and follow up with measurements for three months.

Exclusion Criteria:

* Exclusion criteria include women who have a BMI of over 30 or whom are clinically obese.
* Abdominal obesity can cause low back pain and it increases the lumbosacral angle.
* Women will be excluded who have prior history of back surgery, acute disc herniation, arthritis, immunological disorder, acute fracture and osteoporosis.
* Additional exclusion criteria include high risk pregnancies such as gestational diabetes, preeclampsia, placenta previa and abruptio placentae.
* All of the following could be contributory for low back pain and may affect the biomechanics of the low back.
* If the patients at the NSU clinic have these exclusion criteria documented in their medical chart, they will not be approached for recruitment in the study. During the verbal pre-screening, the research assistant will ask the subject if they have any of the above conditions. If so, they will not be eligible to participate in the study. The same verbal pre-screening will be used at the yoga studio for recruitment. No data will be collected for subjects who are excluded during the pre-screening.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant females in their second or third trimester.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Weight Gain | Every 2-3 weeks in 2nd and/or 3rd trimester for eight weeks
  Amount of weight gain over the 2nd and 3rd trimester in lbs.

SECONDARY OUTCOMES:
Degree of Low Back Pain | Every 2-3 weeks in 2nd and/or 3rd trimester for eight weeks
  Degree of Low Back Pain as measured by the Oswestry Low Back Pain Scale.
Sway Rate | Every 2-3 weeks in 2nd and/or 3rd trimester for eight weeks
  The rate (in mm/s) that subject sways while standing still for 15 seconds.
Deviation of Center of Mass | Every 2-3 weeks in 2nd and/or 3rd trimester for eight weeks
  The degree of weight in percentage and lbs. that shifts anterior or posterior.
Lumbosacral Angle | Every 2-3 weeks in 2nd and/or 3rd trimester for eight weeks
  Degree of lumbosacral angle as measured by an inclinometer.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Wessel, OMS3, Principal Investigator — Nova Southeastern University College of Osteopathic Medicine
Locations (2):
- United States (2):
  - Red Pearl Yoga Studio, Fort Lauderdale, Florida
  - Nova Southeastern University Ob/Gyn Clinic, Fort Lauderdale, Florida